CLINICAL TRIAL: NCT01176929
Title: Effectiveness of Telephone Contact and Professional Coordination for Preventing Recurrent Suicidal Acts
Brief Title: Randomized Controlled and Prospective Trial of a Cohort of People Who Made a Suicide Attempt
Acronym: OSTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OST08017
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Suicide, Attempted
Keywords: Suicide, Attempted; prevention suicidal act; telephone contact; professional coordination
MeSH Terms: conditions — Suicide, Attempted | interventions — National Program of Cancer Registries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional group (Experimental): Usual treatment + prevention program of recurrent suicidal acts
  Interventions: Other: Usual treatment and Prevention program
- Control group (Active Comparator): Usual treatment
  Interventions: Other: Usual Treatment

INTERVENTIONS:
Other: Usual treatment and Prevention program — Prevention program of recurrent suicidal acts includes three interventions:
  * A series of three telephone calls ( the second week , one month and three months after discharge from hospital )
  * A systematic telephone contact with the referring physician
  * A telephone helpline for people who made a suicide attempt and referring physicians.
  Other Names: Prevention program
  Arms: Interventional group
Other: Usual Treatment — Usual Treatment
  Arms: Control group

SUMMARY:
The prevention of recurrent suicidal about people who have made a suicide attempt is a major strand in the prevention of suicide. It is estimated that 10-15 % of people who made a suicide attempt die by suicide. Recidivism rate of suicide increases even faster than the subject is close to the index suicide attempt. A one month recurrence rate is 5 %, 12-25 % at one year. Most people who made a suicide attempt receive ambulatory monitoring. On this population, there is a low adherence to care.

The main objective of the study is to test the effectiveness of a prevention program of recurrent suicidal acts for people who made a suicide attempt.

The secondary objectives of this study are the assessment of adherence to care; the identification of sub - populations benefiting most from this program; the evaluation of the possible generalization level of the program (eligibles persons rate) and its feasibility level.

DETAILED DESCRIPTION:
This is a randomized, controlled and prospective trial comparing an experimental group (usual treatment + interventions) to a control group (usual treatment only). All participants are evaluated after one year of monitoring. The search duration is 2 years (one inclusion year and one year of follow-up). It is planned to include 330 patients, 165 patients in each group.

The program (experimental group) includes three interventions:

* A series of three telephone calls ( the second week , one month and three months after discharge from hospital )
* A systematic telephone contact with the referring physician
* A telephone helpline for people who made a suicide attempt and referring physicians.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years.
* Patients admitted to the emergency department for a suicide attempt.
* Patients referred to outpatient care.
* Patients who have given their written consent.

Exclusion Criteria:

* Patients not affiliated to social security.
* Patients do not have the faculties needed to be evaluated (cognitive or delusional disorder).
* Patients hospitalized for longer than 72 hours.
* Patients can not be recalled by phone (no phone, homeless, incarcerated)
* Patients who do not speak French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
suicidal act frequency | 12 months
  The primary endpoint is the occurrence of a suicidal act (occurrence or not). The suicidal act includes suicide and suicide attempt.

SECONDARY OUTCOMES:
suicide attempts frequency | 12 months
  Number of occurrence of suicide attempts.
Adherence to health care | 12 months
  Adherence to health care:
  Defined by:
  * The Initialization of outpatient care proposed by the suicidology's team at the initial interview or during telephone contacts.
  * The number of consultations within 3 months after the first appointment with the referring doctor.
Number of eligibles persons | 12 months
  Number of eligibles persons:
  Number of people (among all people admitted to the emergency department fo a suicide attempt) meeting the criteria of selection.
Number of participants responding to telephone calls | 12 months
  Number of participants responding to telephone calls:
  We consider the failure to call after three unsuccessful telephone calls to three different days.
Number of people lost sight of | 12 months
  Number of people lost sight of:
  A person is considered lost sight if no information can be obtained after contact with the person himself, a third (nearest designated), a doctor (general practitioner and / or psychiatrist) and the nearest emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud MARCHAND, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris : BICETRE Hospital, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617